CLINICAL TRIAL: NCT01498939
Title: A Single Centre, Randomised, Double-blind, Three-period Cross-over Trial to Investigate the 24-hour Pharmacokinetics After Single Dose of Insulin Detemir in Healthy Chinese Male Subjects
Brief Title: Pharmacokinetics of Insulin Detemir in Healthy Chinese Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN304-1889
Record Dates: First submitted 2011-12-21; First posted 2011-12-26 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin Detemir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- IDet 0.2 U/kg (Experimental)
  Interventions: Drug: insulin detemir
- IDet 0.4 U/kg (Experimental)
  Interventions: Drug: insulin detemir
- IDet 0.8 U/kg (Experimental)
  Interventions: Drug: insulin detemir

INTERVENTIONS:
Drug: insulin detemir — Each subject will be randomly allocated to an insulin detemir dosing sequence. Three doses of insulin detemir (0.2, 0.4 or 0.8 U/kg) will be administered on three inconsecutive days with a wash-out period between each dosing. Injected subcutaneously (s.c., under the skin)

SUMMARY:
This trial is conducted in Asia. The aim of this trial is to investigate the pharmacokinetics after a single dose of insulin detemir in healthy Chinese male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 18 and 25 kg/m^2 (both inclusive)
* Fasting plasma glucose maximum 6 mmol/L
* Non-smoker
* Considered generally healthy upon completion of medical history, physical examination and laboratory assessments, as judged by the Investigator

Exclusion Criteria:

* Known or suspected allergy to trial product(s) or related products
* Previous participation in this trial. Participation is defined as randomisation
* Receipt of any investigational drug within the last three months prior to this trial
* History of alcohol or drug abuse

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2007-08; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Area under the insulin detemir concentration curve | from time zero to 24 hour

SECONDARY OUTCOMES:
Area under the insulin detemir concentration curve
Maximum serum insulin detemir concentration
Time to maximum serum insulin detemir concentration
Mean residence time (MRT)
Terminal half-life
Insulin detemir clearance
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Beijing, Beijing Municipality, China

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com